CLINICAL TRIAL: NCT01220973
Title: Phase II Trial of Atorvastatin and Celecoxib in Patients With Hormone-Dependent Prostate-Specific Antigen Progression After Local Therapy for Prostate Cancer.
Brief Title: Atorvastatin Calcium and Celecoxib in Treating Patients With Rising PSA Levels After Local Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Goodin, PharmD, Professor of Medicine, RWJMS, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0220090006, 080811; 0220090006 (Other: IRB number); NCI-2012-00540 (Other: CTRP (Clinical Trails Reporting Program))
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; stage III prostate cancer; recurrent prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Atorvastatin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin and Celecoxib (Experimental)
  Interventions: Drug: atorvastatin calcium; Drug: celecoxib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: atorvastatin calcium
Drug: celecoxib
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Atorvastatin calcium and celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving atorvastatin calcium together with celecoxib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving atorvastatin calcium together with celecoxib works in treating patients with rising PSA levels after local therapy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the effect on the biological activity, as assessed by prostate-specific antigen (PSA) response, of atorvastatin calcium and celecoxib in patients with D0 prostate cancer.

Secondary

* To document the safety and feasibility of atorvastatin calcium and celecoxib in patients with early-stage prostate cancer.
* To evaluate the effects of the combination of atorvastatin calcium and celecoxib on nuclear factor-kB (NFkB), extracellular signal-regulated kinase (ERK), prostaglandin E2 (PGE2), and IL6 in peripheral blood mononuclear cells (PBMC).

OUTLINE: This is a multicenter study.

Patients receive oral atorvastatin calcium once daily and oral celecoxib twice daily on days 1-28. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood sample collection at baseline and after completion of study therapy for correlative studies.

After completion of study therapy, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * Stage D0 disease

    * Tumor originally diagnosed as being limited to the prostate and now having a rising prostate-specific antigen (PSA) after definitive local therapy
* Must have undergone local treatment via prostatectomy or radiotherapy

  * PSA values must be ≥ 0.2 ng/mL as determined by 2 measurements, ≥ 1 month apart and ≥ 6 months after prostatectomy
  * PSA values must be ≥ 2.0 ng/mL as determined by 2 measurements, ≥ 1 month apart and ≥ 6 months after radiotherapy
  * The first two PSA values along with a third value must all be rising (i.e., there must be an overall rising trajectory, such that the third value cannot be lower than the first value)
* No metastatic disease by baseline bone scan and CT scan of the abdomen and/or pelvis

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* ECOG performance status 0-2
* WBC ≥ 3,500/µL
* ANC ≥ 1,500/µL
* Platelet count > 100,000/µL
* Hemoglobin > 10 g/dL
* Serum creatinine < 1.5 mg/dL OR creatinine clearance > 50 mL/min
* Total bilirubin normal
* SGOT and/or SGPT normal
* No serious concomitant systemic disorder that, at the discretion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* No second primary malignancy within the past 5 years except adequately treated in situ carcinoma (e.g., non-melanomatous carcinoma of the skin) or other malignancy with no evidence of recurrence
* No active clinically significant infection requiring antibiotics
* No history of coronary artery disease
* No myocardial infarction within the past 6 months
* No sulfa allergy
* No history of gastrointestinal bleeding

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hormone-ablative treatment

  * Prior neoadjuvant hormone-ablative therapy allowed provided it was completed ≥ 3 months ago
* More than 4 weeks since prior herbal products with hormonal activity such as soy, saw palmetto, or PC-SPES
* No prior or concurrent nonsteroidal anti-inflammatory drug (NSAIDS) for 7 consecutive days
* No COX-2 inhibitor and/or statin within the past 6 months
* No concurrent warfarin or any other anticoagulant, calcitriol, fibric acid derivatives, lipid-modifying doses of niacin, or strong cytochrome P450 3A4 inhibitors (e.g., cyclosporine, erythromycin, clarithromycin, and azole antifungals) or inducers (e.g., St John wort)
* No other concurrent anticancer agents or therapies including chemotherapy, hormonal therapy, radiotherapy, or experimental therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-02; Primary Completion 2014-11-18 (Actual); Study Completion 2014-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Goodin, PhD, FCCP, BCOP, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (4):
- United States (4):
  - Karmanos Cancer Center, Detroit, Michigan
  - Cooper Hospital, Camden, New Jersey
  - Robert Wood Johnson University Hospital at Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey Oncology Group. The study was open to accrual on 02/25/2009 and closed to accrual on 11/13/2012.
Pre-assignment Details: We are reporting results on 27 eligible patients. Seven patients were deemed ineligible.
Groups:
- Atorvastatin and Celecoxib: atorvastatin calcium
  celecoxib
  laboratory biomarker analysis
Period: Overall Study
Arm/Group | Atorvastatin and Celecoxib
Started | 27
Completed | 23
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin and Celecoxib
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: PSA Response
Description: PSA response was defined as a decrease in slope of at least 25%, when log (PSA) is plotted vs. time.
Time Frame: 6 months
Population: A total of 27 patients were enrolled but only 26 were evaluable as one patient withdrew consent prior to starting therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin and Celecoxib
Number analyzed (Participants) | 26
Participants | 14
Statistical Analysis 1: Comparison: Atorvastatin and Celecoxib; Test type: Other; Slope = 0.74

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 900 days per patient.
Arm/Group | Atorvastatin and Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes